CLINICAL TRIAL: NCT03643419
Title: Clinical Study of Treatment of Acute Spinal Cord Injury by Near Infrared Light Irradiation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20172036-1
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injuries; Photobiology; Neurological Rehabilitation; Near Infrared Light Irradiation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Laminectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminectomy (Sham Comparator)
  Interventions: Procedure: Laminectomy
- Laminectomy & Irradiation (Experimental)
  Interventions: Procedure: Laminectomy; Device: Spinal nerve laser therapeutic apparatus（Composed of 808-band fully automatic control laser device and implantable 360° scattering medical fiber）

INTERVENTIONS:
Procedure: Laminectomy — According to the standard procedure of laminectomy for acute spinal cord injury
Device: Spinal nerve laser therapeutic apparatus（Composed of 808-band fully automatic control laser device and implantable 360° scattering medical fiber） — According to the standard procedure of decompression of laminectomy for acute spinal cord injury, the patient in the Near Infrared Light Irradiation Group placed the implantable 360° scattering fiber laterally above the operation area at the end of the operation. Near infrared light irradiation is applied by spinal nerve laser therapeutic apparatus every day from the day after surgery, once a day for 60 minutes each time.
  Arms: Laminectomy & Irradiation

SUMMARY:
The purpose of this study was to observe the therapeutic effect of near-infrared light irradiation on the treatment of acute spinal cord injury in humans, and whether it can promote the recovery of neurological function. Half of the patients underwent laminectomy and decompression surgery, and the other half of the patients were implanted with irradiated fibers for irradiation after surgery.

DETAILED DESCRIPTION:
The annual incidence of spinal cord injury has increased year by year, and there is currently no effective treatment.

Near-infrared light has been widely used in clinical medicine because of its bio-stimulating effect, convenient use, harmless to the body, easy to be accepted by patients, and convenient for clinical promotion. The near-infrared light biostimulation effect can enhance the activity of various enzymes, inhibit inflammatory cells, inhibit neuronal apoptosis, and promote nerve regeneration. It has been widely confirmed and widely used in the rehabilitation of central nervous system and peripheral nerve injury. However, the position of the spinal cord is deep, and the depth of illumination used by laser treatment equipment is generally difficult to reach.

The implantable 360° scattering fiber the investigators developed was implanted in the surgical site together with the drainage tube for irradiation treatment without additional patient damage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as acute spinal cord injury (ASIA grade A-C) (thoracic segment) requiring surgical laminectomy
* The patient determined by the investigator to be eligible for the illuminating fiber implanted in this clinical trial
* The patient fully understands the content and requirements of this clinical trial and is able to complete the follow-up according to the time specified in the protocol
* Voluntary participation in clinical validation and signing informed consent

Exclusion Criteria:

* The patient has a systemic infection or a local infection at the target surgical site
* The patient has more than 2 segments of spinal cord injury, and the vital signs are unstable
* A patient with a malignant tumor that does not involve the target surgical site
* Patient life expectancy is less than one year
* Pregnant or lactating women
* The patient is too obese, BMI ≥ 40
* Patients with other systemic diseases who are using corticosteroids, or patients with growth factors, or long-term use of non-steroidal anti-inflammatory drugs
* Patients have a history of endocrine diseases affecting bone metabolism (such as diabetes, metabolic bone disease, etc.) or autoimmune diseases (such as multiple sclerosis)
* Alcohol abuse within one year (average daily alcohol consumption > 40g, equivalent to 50ml alcohol 50ml, or smoking ≥ 40 / day, or drug abusers)
* Participating in other drug or device clinical trials

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline ASIA Rating Scale at 6 Months | 6 Months
  The ASIA rating scale was used to evaluate the patient's function, and the scores of each major item were obtained according to the weighting factors of each major item, with a total score of 0 to 100 points.
Change from Baseline ASIA Rating Scale at 12 Months | 12 Months
  The ASIA rating scale was used to evaluate the patient's function, and the scores of each major item were obtained according to the weighting factors of each major item, with a total score of 0 to 100 points.
Change from Baseline EMG at 6 Months | 6 Months
  The motor evoked potentials（MEP) and sensory evoked potentials(SEP) were evaluated, and the differences in the latency of the evoked potential N1 wave between the two groups were compared.
Change from Baseline EMG at 12 Months | 12 Months
  The motor evoked potentials（MEP) and sensory evoked potentials(SEP) were evaluated, and the differences in the latency of the evoked potential N1 wave between the two groups were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Wang, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sekhon LH, Fehlings MG. Epidemiology, demographics, and pathophysiology of acute spinal cord injury. Spine (Phila Pa 1976). 2001 Dec 15;26(24 Suppl):S2-12. doi: 10.1097/00007632-200112151-00002. PMID 11805601
- [Background] Khan I, Tang E, Arany P. Molecular pathway of near-infrared laser phototoxicity involves ATF-4 orchestrated ER stress. Sci Rep. 2015 Jun 1;5:10581. doi: 10.1038/srep10581. PMID 26030745
- [Background] Black B, Vishwakarma V, Dhakal K, Bhattarai S, Pradhan P, Jain A, Kim YT, Mohanty S. Spatial temperature gradients guide axonal outgrowth. Sci Rep. 2016 Jul 27;6:29876. doi: 10.1038/srep29876. PMID 27460512
- [Background] Chen YJ, Wang YH, Wang CZ, Ho ML, Kuo PL, Huang MH, Chen CH. Effect of low level laser therapy on chronic compression of the dorsal root ganglion. PLoS One. 2014 Mar 4;9(3):e89894. doi: 10.1371/journal.pone.0089894. eCollection 2014. PMID 24594641